CLINICAL TRIAL: NCT02715505
Title: A Single-arm, Open-label, Study to Evaluate the Safety and Exploratory Efficacy of HSC835 in Patients With Inherited Metabolic Disorders (IMD) Undergoing Stem Cell Transplantation After Reduced Intensity Conditioning
Brief Title: Safety and Exploratory Efficacy of HSC835 in Patients With Inherited Metabolic Disorders (IMD)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was cancelled with no patients
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHSC835X2203
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Inherited Metabolic Disorders IMD
Keywords: Hurler syndrome, MLD, Krabbe, cALD, Hematopoietic Stem Cell Transplantation (HSCT)
MeSH Terms: conditions — Mucopolysaccharidosis I; Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HSC835 (Experimental): HSC835 is an expanded umbilical cord blood product used during single umbilical cord blood transplantation
  Interventions: Drug: Umbilical cord blood transplantation with HSC835

INTERVENTIONS:
Drug: Umbilical cord blood transplantation with HSC835 — Hematopoietic Stem cell transplantation will be done with the cell therapy product HSC835
  Other Names: Spanlecortemlocel

SUMMARY:
This study is designed to assess the safety and exploratory efficacy of using HSC835 in patients with Inherited Metabolic Disorders (IMD) undergoing stem cell transplantation.

DETAILED DESCRIPTION:
This phase II study is designed to assess the safety of the Novartis product HSC835 and its ability to achieve donor blood stem cell engraftment in patients with certain Inherited Metabolic Disorders who undergo stem cell transplantation. A reduced intensity conditioning will be used prior to transplantation. Patients with Hurler syndrome, MLD, Krabbe or cALD could be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hurler syndrome, Metachromatic leukodystrophy (MLD), Globoid cell leukodystrophy (Krabbe) or Cerebral adrenoleukodystropy (cALD) -Adequate organ function -Availability of eligible donor material

Exclusion Criteria:

* Availability of a matched-related donor who is not a carrier of the same genetic defect -Active infection at screening -Prior myeloablative transplant -Pregnant or nursing women and women of child bearing potential unless using highly effective contraception methods. For the pediatric population, female patients of child bearing potential who do not agree to abstinence or agree to use highly effective contraception methods -Sexually active male patients unless using condoms as contraception -Human Immunodeficiency virus (HIV) infection

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-10 (Estimated); Primary Completion 2020-05-18 (Estimated); Study Completion 2020-05-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of infusional toxicities | 48 hours
Incidence of neutrophil recovery | 42 days
Incidence of graft failure | 42 days

SECONDARY OUTCOMES:
Time to neutrophil recovery | 42 days
Time to platelet recovery | 180 days
Number of patients with grade II-IV acute graft versus host disease (aGVHD) | 100 days
Number of patients with chronic graft versus host disease (cGVHD) | 1 and 2 years
Incidence of death | 100 days, 1 year and 2 years

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com